CLINICAL TRIAL: NCT00484068
Title: Effect of Chicken-Based Diet Versus Enalapril on Albuminuria in Patients With Type 2 Diabetes and Microalbuminuria: a One-Year Randomized Controlled Study
Brief Title: Chicken-Diet vs. Enalapril to Reduce Albuminuria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCPA-98238
Record Dates: First submitted 2007-06-06; First posted 2007-06-08 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-06

CONDITIONS: Microalbuminuria; Diabetic Nephropathy
Keywords: type 2 diabetes; microalbuminuria; chicken-based diet; ACE inhibitor
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — Enalapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: enalapril
Procedure: chicken diet

SUMMARY:
Diabetic nephropathy (DN) is a chronic diabetic complication and affects up to 40% of patients. The first line treatment for DN is angiotensin blockers drugs that are used to reduce the protein concentration in urine.Previous data showed that this protein, namely albuminuria, could also be reduced in a short term-period by the replacement of red meat in the diet with chicken. The aim of this study is to compare the effects of this chicken diet with enalapril on albuminuria in a long-term period( 12 months)in type 2 diabetic patients.

DETAILED DESCRIPTION:
Replacement of red meat in the diet with chicken reduces urinary albumin excretion rate (UAER) and improves lipid profile in type 2 diabetic patients with micro- and macroalbuminuria in short term studies. The aim of this study was to compare the long-term effect of a chicken-based diet (CD) versus enalapril treatment on renal function and lipid profile in microalbuminuric type 2 diabetic patients. In this 12-month controlled clinical trial 28 patients were randomized to an experimental diet (CD plus active placebo) or enalapril treatment (enalapril 10 mg/day plus patient's usual diet). UAER (immunoturbidimetry), blood pressure levels, anthropometric indices, and compliance with the diet were evaluated monthly. Glomerular filtration rate (51Cr-EDTA), lipid, glycemic, and nutritional indices were measured at baseline, and quarterly. UAER was reduced after CD [n=13; 62.8 (38.4-125.1) to 49.1 (6.2-146.5) mcg/min; P<0.001] and after enalapril treatment [n=15; 55.8 (22.6-194.3) to 23.1 (4.0-104.9) mcg/min; P<0.001]. The reduction of UAER was already significant at 4th month, and there was no difference between the UAER reduction after CD [32% (95% CI: 6.7-57.6) and after enalapril treatment [44.7% (95% CI: 28.3-61.1); P=0.366]. In conclusion, CD and the ACE inhibitor enalapril promoted similar UAER reduction in patients with type 2 diabetes and microalbuminuria. A chicken-based diet might represent an additional therapeutic approach to management of diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus (according to World Health Organization criteria) attending the Endocrine Division's outpatient clinic at Hospital de Clínicas de Porto Alegre, Brazil. Patients were selected according to the following criteria: age <75 years, A1c <10%, 24-hour UAER 20 mcg/min and 199 mcg/min confirmed at least twice in a 6-month period, serum triglycerides <400 mg/dl and normal liver and thyroid function tests.

Exclusion Criteria:

* Patients were excluded from the study if they had BMI >34 kg/m2, serum creatinine >1.5 mg/dl, repeated episodes of urinary tract infection, other renal diseases, symptomatic autonomic neuropathy, heart failure, and acute myocardial infarction, coronary artery revascularization procedures or stroke within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-01; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
urinary albumin excretion | during study
serum lipids | during study
nutritional status | during study

CONTACTS AND LOCATIONS:
Overall Officials: Jorge L Gross, MD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- HCPortoAlegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Result] Gross JL, Zelmanovitz T, Moulin CC, De Mello V, Perassolo M, Leitao C, Hoefel A, Paggi A, Azevedo MJ. Effect of a chicken-based diet on renal function and lipid profile in patients with type 2 diabetes: a randomized crossover trial. Diabetes Care. 2002 Apr;25(4):645-51. doi: 10.2337/diacare.25.4.645. PMID 11919119
- [Result] de Mello VD, Zelmanovitz T, Perassolo MS, Azevedo MJ, Gross JL. Withdrawal of red meat from the usual diet reduces albuminuria and improves serum fatty acid profile in type 2 diabetes patients with macroalbuminuria. Am J Clin Nutr. 2006 May;83(5):1032-8. doi: 10.1093/ajcn/83.5.1032. PMID 16685043